CLINICAL TRIAL: NCT01013285
Title: Phase II Trial of Bevacizumab in Combination With Temozolomide and Regional Radiation Therapy for Upfront Treatment of Patients With Newly-diagnosed Glioblastoma Multiforme
Brief Title: Bevacizumab, Temozolomide, and External Beam Radiation Therapy as First-Line Therapy in Treating Patients With Newly Diagnosed Glioblastoma Multiforme or Gliosarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-000558; UCLA-0604016; AVF3770s; CDR0000628787; GENENTECH-UCLA-0604016
Record Dates: First submitted 2009-11-11; First posted 2009-11-13 (Estimated); Results first posted 2020-09-21 (Actual); Last update posted 2020-09-21 (Actual); Status verified 2016-04

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult giant cell glioblastoma; adult gliosarcoma; adult glioblastoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Glioblastoma; Gliosarcoma | interventions — Bevacizumab; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- bevacizumab, temozolomide, external beam radiation (Experimental)
  Interventions: Biological: bevacizumab; Drug: temozolomide; Radiation: external beam radiation therapy

INTERVENTIONS:
Biological: bevacizumab
Drug: temozolomide
Radiation: external beam radiation therapy

SUMMARY:
RATIONALE: Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Bevacizumab may also stop the growth of tumor cells by blocking blood flow to the tumor. Drugs used in chemotherapy, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high energy x-rays to kill tumor cells. Giving bevacizumab together with temozolomide and radiation therapy may kill more tumor cells.

PURPOSE: This phase II trial is studying the side effects and how well giving bevacizumab together with temozolomide and external beam radiation therapy works when given as first-line therapy in treating patients with newly diagnosed glioblastoma multiforme or gliosarcoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To investigate the safety and tolerability of bevacizumab in combination with temozolomide and external beam fractionated regional radiotherapy as first-line treatment in patients with newly diagnosed glioblastoma multiforme or gliosarcoma. (Pilot phase)
* To estimate the overall survival of patients treated with this regimen. (Expansion phase)

Secondary

* To further investigate the safety and tolerability of this regimen in these patients. (Expansion phase)
* To isolate DNA, RNA, and protein from frozen and paraffin-embedded archival tumor samples for evaluations, such as immunohistochemical pathway profiling of vascular endothelial growth factor (VEGF)-dependent angiogenic pathways, gene expression microarray, and O-6 methylguanine DNA methyltransferase (MGMT) promoter methylation status to define important molecular features of treatment response.

OUTLINE: This is a multicenter study.

Patients undergo external beam fractionated regional radiotherapy once daily 5 days a week for 6 weeks and receive concurrent oral temozolomide once daily for 6 weeks. Patients also receive bevacizumab IV over 30-90 minutes every 2 weeks beginning on the first day of radiotherapy and continuing in the absence of disease progression or unacceptable toxicity. Beginning 2-5 weeks after completion of radiotherapy, patients receive oral temozolomide on days 1-5. Treatment with temozolomide repeats every 28 days for up to 24 courses in the absence of disease progression or unacceptable toxicity.

Blood and frozen and paraffin-embedded tumor tissue samples are collected for biomarker and genetic analysis.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed intracranial glioblastoma multiforme (GBM) or gliosarcoma.
* Prior histologic diagnosis of low-grade glioma allowed provided it has been upgraded to GBM after repeat resection
* Has undergone surgery to collect tumor tissue 3-6 weeks ago
* Measurable or assessable disease is not required
* Karnofsky performance status 60-100%
* Life expectancy > 8 weeks
* White Blood Cell (WBC) ≥ 3,000/mm³
* Absolute Neutrophil Count (ANC) ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 10 g/dL (transfusion allowed)
* Serum Glutamate Oxaloacetate Transaminase (SGOT) < 2.5 times upper limit of normal (ULN)
* Bilirubin < 2.5 times ULN
* INR (international normalized ratio) ≤ 1.5 times ULN (except if on therapeutic anticoagulation therapy)
* aPTT (activated partial thromboplastin time) ≤ 1.5 times ULN (except if on therapeutic anticoagulation therapy)
* Creatinine < 1.5 mg/dL
* Urine protein:creatinine ratio < 1.0
* Negative pregnancy test
* Fertile patients must use effective contraception
* More than 28 days since prior major surgical procedures or open biopsy (other than craniotomy)
* More than 7 days since prior minor surgical procedures (e.g., placement of PortoCath (port-a-cath - a port placed under the subjects skin), stereotactic biopsy, fine-needle aspirations, or core biopsies)
* More than 4 weeks since prior and no concurrent participation in another experimental drug study.
* Prior or concurrent corticosteroids, anti-epileptic drugs, analgesics, or other drugs to treat symptoms or prevent complications are allowed
* Concurrent full-dose warfarin or its equivalent (i.e., unfractionated and/or low molecular weight heparin) allowed

Exclusion Criteria:

* unstable angina
* BP > 150/100 mm Hg
* New York Heart Association (NYHA) class II-IV congestive heart failure
* myocardial infarction within the past 6 months
* stroke within the past 6 months
* clinically significant peripheral vascular disease
* evidence of bleeding diathesis or coagulopathy
* intracerebral abscess within past 6 months
* abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within the past 6 months
* serious, non-healing wound, ulcer, or bone fracture
* Any wound requiring surgical intervention (including scalp wounds requiring cranioplasty) allowed provided the wound is clean and without further infection post-surgical intervention
* significant traumatic injury within the past 28 days
* concurrent serious uncontrolled medical illness including, but not limited to, the following:
* Ongoing or active infection requiring IV antibiotics
* Psychiatric illness/social situation that would limit compliance with study requirements
* Disorders associated with significant immunocompromised state (e.g., HIV, systemic lupus erythematosus)
* other cancer within the past 3 years, except nonmelanoma skin cancer or carcinoma in situ of the cervix
* disease that would obscure toxicity or dangerously alter drug metabolism
* significant medical illness that, in the investigator's opinion, cannot be adequately controlled with appropriate therapy or would compromise the patient's ability to tolerate study therapy
* prior radiotherapy to the brain
* prior cytotoxic or non-cytotoxic drug therapy or experimental drug therapy for the brain tumor
* prior Gliadel wafers
* concurrent participation in any other clinical trial
* concurrent GM-CSF (granulocyte-macrophage colony-stimulating factor)
* concurrent stereotactic radiosurgery or brachytherapy
* concurrent major surgical procedure
* other concurrent anticancer therapy, including chemotherapy, hormonal therapy, radiotherapy, or immunotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2006-06; Primary Completion 2013-10 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Albert Lai, MD, Principal Investigator — Ronald Reagan University of California, Los Angeles (UCLA) Medical Center
Locations (1):
- Jonsson Comprehensive Cancer Center, University of California, Los Angeles (UCLA), Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Seventy patients with newly diagnosed Glioblastoma Multiforme were enrolled between August 2006 and November 2008 from two participating sites, comprised of University of California, Los Angeles (UCLA) and Kaiser Permanente Los Angeles.
Pre-assignment Details: Control cohort was derived from University of California, Los Angeles/Kaiser Permanente Los Angeles patients treated with first-line radiation therapy and temozolomide who had mostly received bevacizumab at recurrence.
Groups:
- Treatment Arm: bevacizumab
  temozolomide
  external beam radiation therapy
- Historical Control UCLA/KPLA: A University of California, Los Angeles/Kaiser Permanente Los Angeles(KPLA) control cohort of newly diagnosed patients treated with first-line radiation therapy and temozolomide who had mostly received bevacizumab at recurrence was derived for comparison.
Period: Overall Study
Arm/Group | Treatment Arm | Historical Control UCLA/KPLA
Started | 70 | 110
Completed | 22 | 21
Not Completed | 48 | 89
Not completed — Death | 48 | 89

BASELINE CHARACTERISTICS:
Groups:
- Historical Control UCLA/Kaiser: A University of California, Los Angeles/Kaiser Permanente Los Angeles(KPLA) control cohort of newly diagnosed patients treated with first-line radiation therapy and temozolomide who had mostly received bevacizumab at recurrence was derived for comparison. Data excluded where records not complete
- Total: Total of all reporting groups
Arm/Group | Treatment Arm | Historical Control UCLA/Kaiser | Total
Number analyzed (Participants) | 70 | 110 | 180
Age, Continuous [Median (Full Range); unit: years] | 57.4 [31.3 to 75.8] | 59.4 [20.5 to 90] | 59.305 [20.5 to 90]
Age, Customized [Number; unit: participants]
  < 50 years | 15 | 30 | 45
  >= 50 years | 55 | 80 | 135
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 40 | 71
  Male | 39 | 70 | 109
Enrollment by Site [Number; unit: participants]
  UCLA | 38 | 61 | 99
  KPLA | 32 | 49 | 81
Karnofsky performance status [Number; unit: participants] — Karnofsky performance status:
  100: Normal no complaints; no evidence of disease. 90: Able to carry on normal activity; minor signs or symptoms of disease. 80: Normal activity with effort; some signs or symptoms of disease. 70: Cares for self; unable to carry on normal activity or to do active work. 60: Requires occasional assistance, but is able to care for most of his personal needs. 100 best, the lower the number the worse outcome.
  participants
    100 | 8 | 13 | 21
    90 | 27 | 62 | 89
    80 | 27 | 23 | 50
    70 | 5 | 8 | 13
    60 | 3 | 4 | 7
Extent of surgery [Number; unit: participants]
  Biopsy | 2 | 23 | 25
  Subtotal resection | 40 | 40 | 80
  Gross total resection | 28 | 47 | 75
Recursive partitioning analysis by class [Number; unit: participants] — According to a 2003 study, glioblastoma multiforme prognosis can be divided into three subgroups dependent on Karnofsky Performance Status (KPS), the age of the patient, and treatment.
  MST= Median Survival Time in months. III: Age < 50, KPS ≥ 90; IV: Age < 50, KPS < 90, Age ≥ 50, KPS ≥ 70, surgical removal, good neurologic function;
  V + VI, Age ≥ 50, KPS ≥ 70, surgical removal with poor neurologic function:
  Age ≥ 50, KPS ≥ 70, no surgical removal. Age ≥ 50, KPS < 70
  participants
    III: MST 17.1 | 9 | 27 | 36
    IV: MST 11.2 | 32 | 45 | 77
    V: MST 7.5 | 29 | 37 | 66
    VI: MST 7.5 | 0 | 1 | 1
Follow-up [Median (Full Range); unit: years] | 24.2 [12 to 40] | 41.8 [29 to 58] | 36.616 [12 to 58]
Deaths [Number; unit: participants] | 48 | 89 | 137
Recurrent treatment [Number; unit: participants]
  Progressed | 56 | 96 | 152
  Progressed with chemotherapy | 39 | 64 | 103
  Progressed with bevacizumab | 29 | 57 | 86
MGMT (O-6-Methylguanine-DNA Methyltransferase) promoter methylation [Number; unit: participants] — The MGMT (O-6-Methylguanine-DNA Methyltransferase) promoter methylation status was not available for all of the historical control samples. Therefore, only the samples with the information available were included.
  participants
    Methylated | 29 | 28 | 57
    Unmethylated | 41 | 43 | 84
IDH1 (Isocitrate dehydrogenase 1 ) mutational status [Number; unit: participants] — [1] The IDH1 (Isocitrate dehydrogenase 1 ) promoter methylation status was not available for all of the historical control samples. Therefore, only the samples with the information available were included.
  participants
    Wild type | 65 | 68 | 133
    IDH1-R132H mutation | 5 | 3 | 8

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Time Frame: 2 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment Arm | Historical Control UCLA/KPLA
Number analyzed (Participants) | 70 | 110
Months | 19.6 [16.1 to 23.3] | 21.1 [18.9 to 25.2]

2. Secondary Outcome: Time to Disease Progression
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: 2 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment Arm | Historical Control UCLA/KPLA
Number analyzed (Participants) | 70 | 110
Months | 13.6 [11.1 to 16.5] | 7.6 [5.9 to 10.8]

3. Secondary Outcome: Progression-free Survival at 6 Months
Description: participants who were alive and disease progression free at 6 months
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment Arm | Historical Control UCLA/KPLA
Number analyzed (Participants) | 70 | 110
percentage of participants | 88.4 [81.17 to 96.3] | 58.3 [49.7 to 68.4]

4. Secondary Outcome: Radiographic Response (When Evaluable)
Description: Radiation therapy (RT) median from diagnosis to RT. Patients will have brain MRI evaluation of response and progression every 8 weeks starting from the day 56 scan obtained 2 weeks after completion of radiation and daily temozolomide and assessment will be conducted on a 7-point scale. This scale is expected to be more useful in this study because many newly-diagnosed patients are likely not to have evaluable disease due to gross total resections. Determination of whether progression occurs based on the day 56 scan will take into account the untreated window between baseline MRI and day of 1 of study.
  7 Point Likert Scale: 3 to -3, 3 means complete resolution of tumor, and -3 means new lesion. A -2 or -3 assessment will be taken as tumor progression.
  complete resolution of tumor: 3
  tumor resolved 3 tumor definitely smaller: 2 tumor probably smaller: 1 tumor unchanged: 0 tumor probably worse: -1 tumor definitely worse: -2 New Lesion: -3
Time Frame: 2 years
Measure: Median (90% Confidence Interval); unit: Weeks
Arm/Group | Treatment Arm | Historical Control UCLA/KPLA
Number analyzed (Participants) | 70 | 110
Weeks | 4.14 [3 to 6.9] | 5 [1.7 to 10.7]

5. Secondary Outcome: Median Overall Survival (OS) Based on the MGMT Promoter Methylation Status
Description: IDH1 and MGMT methylation are important independent prognostic biomarkers that have to be included in a Cox regression model. In addition, subgroup analysis could reveal differential sensitivities to the treatment arm. The MGMT promoter methylation status, IDH1 mutation status were not available for all of the control samples. Therefore, only the samples with both info available were included in the analysis. Baseline analysis results are included in the Baseline Characteristics module.
Time Frame: 2 years
Population: Description: Kaplan-Meier analysis of overall survival was performed.
Measure: Median (Full Range); unit: months
Arm/Group | Treatment Arm | Historical Control UCLA/KPLA
Number analyzed (Participants) | 70 | 71
months
  Median Overall survival of MGMT Methylated | 24.7 [11.7 to 38.2] | 26.7 [3.5 to 43.2]
  Median Overall survival of MGMT Unmethylated | 15.9 [5.7 to 31.5] | 18.2 [2.1 to 48.1]

ADVERSE EVENTS:
Time Frame: Data collected through study completion, 2.25 years.
Description: period coinciding with Aug 23, 2006 - Nov 26, 2008
Groups:
- Bevacizumab, Temozolomide, External Beam Radiation: bevacizumab
  temozolomide
  external beam radiation therapy
Arm/Group | Bevacizumab, Temozolomide, External Beam Radiation
Serious Adverse Events (participants affected / at risk) | 54/70
Other Adverse Events (participants affected / at risk) | 14/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab, Temozolomide, External Beam Radiation (N=70)
Acute dehydration (General disorders) | 1 (1)
Acute inferior wall MI (Gastrointestinal disorders) | 1 (1)
Acute renal failure (Renal and urinary disorders) | 1 (1)
Altered mental status (Psychiatric disorders) | 6 (7)
Bowel perforation (Gastrointestinal disorders) | 1 (1)
Coma (General disorders) | 1 (1)
congestive heart failure (Cardiac disorders) | 1 (1)
Craniotomy wound w/cerebrospinal fluid leak (Investigations) | 2 (2)
Deep vein thrombosis (Vascular disorders) | 2 (2)
Falling episode/syncopal episode status post fall (Ear and labyrinth disorders) | 1 (1)
Fatigue (General disorders) | 2 (2)
Flu like symptoms (General disorders) | 1 (1)
Fungal infection (Left lung) (Infections and infestations) | 1 (1)
Gastroenteritis due to E. coli. (Gastrointestinal disorders) | 1 (1)
GI Bleeding (Gastrointestinal disorders) | 2 (2)
Hypertension (General disorders) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
hypotention (General disorders) | 1 (1)
Left retinal detachment (Eye disorders) | 1 (1)
leukopenia (Blood and lymphatic system disorders) | 1 (2)
Nausea (Gastrointestinal disorders) | 2 (2)
Nephritic proteinuria (Blood and lymphatic system disorders) | 1 (1)
Nephrotic syndrome (Blood and lymphatic system disorders) | 1 (1)
neutropenia (Blood and lymphatic system disorders) | 1 (2)
obstructive uropathy (Renal and urinary disorders) | 1 (1)
Perforated sigmoid diverticulum (Gastrointestinal disorders) | 1 (1)
pulmonary embolism (Cardiac disorders) | 4 (4)
Renal failure (Renal and urinary disorders) | 1 (2)
Seizure (Nervous system disorders) | 3 (3)
Steroid-induced psychosis (Psychiatric disorders) | 1 (1)
Stroke (Blood and lymphatic system disorders) | 1 (1)
thrombocytopenia (Blood and lymphatic system disorders) | 1 (2)
Transient Ischemic Attack (Blood and lymphatic system disorders) | 1 (1)
Upper Resp. tract Infection (Infections and infestations) | 1 (1)
Urinary Tract Infection (Renal and urinary disorders) | 1 (2)
Ventriculoperitoneal shunt placement. (Cardiac disorders) | 1 (1)
Wound dehisicence of frontal wound (Musculoskeletal and connective tissue disorders) | 1 (1)
Wound infection (Infections and infestations) | 1 (1)
vomiting (Gastrointestinal disorders) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab, Temozolomide, External Beam Radiation (N=70)
Fatigue (General disorders) | 12 (12)
Hypertension (Blood and lymphatic system disorders) | 7 (7)
Proteinuria (Blood and lymphatic system disorders) | 5 (5)
Syncope (General disorders) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No